CLINICAL TRIAL: NCT06360640
Title: A First-in-human, Randomised, Double-blind, Placebo-controlled, Single Ascending Dose Trial to Evaluate Safety, Tolerability, and Pharmacokinetics of APC148 in Healthy Adults
Brief Title: A First-in-human Trial to Evaluate Safety, Tolerability, and Pharmacokinetics of APC148 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AdjuTec Pharma AS (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: APC148-001; 2023-507939-38-00 (Other: EU Trial no)
Record Dates: First submitted 2024-03-05; First posted 2024-04-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, 6 sequential cohorts.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- 50 mg of APC148 and placebo (Experimental): Cohort 1: 4 participants receives 3 hours IV administration of 50 mg APC148, and 2 participants placebo.
  Interventions: Drug: APC148 and Placebo
- 150 mg of APC148 and placebo (Experimental): Cohort 2: 6 participants receives 3 hours IV administration of 150 mg APC148 and 2 participants placebo.
  Interventions: Drug: APC148 and Placebo
- 300 mg of APC148 and placebo (Experimental): Cohort 3: 6 participants receives 3 hours IV administration of 300 mg APC148 and 2 participants placebo.
  Interventions: Drug: APC148 and Placebo
- 450 mg of APC148 and placebo (Experimental): Cohort 4: 6 participants receives 3 hours IV administration of 450 mg APC148 and 2 participants placebo.
  Interventions: Drug: APC148 and Placebo
- 600 mg of APC148 and placebo (Experimental): Cohort 5: 6 participants receives 3 hours IV administration of 600 mg APC148 and 2 participants placebo.
  Interventions: Drug: APC148 and Placebo
- 900 mg of APC148 and placebo (Experimental): Cohort 6: 6 participants receives 3 hours IV administration of 900 mg APC148 and 2 participants placebo.
  Interventions: Drug: APC148 and Placebo

INTERVENTIONS:
Drug: APC148 and Placebo — IV infusion

SUMMARY:
The purpose of this first-in-human trial is to investigate the safety, tolerability, and pharmacokinetics of APC148 after intravenous (IV) infusion of single ascending doses in healthy adults.

DETAILED DESCRIPTION:
Participants will receive a single 3-hours IV infusion of APC148 or placebo. 6 sequential cohorts are planned. The first 2 subjects in each cohort will be dosed in a sentinel fashion. The subjects will be followed for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent for participation in the trial.
* Healthy females of non-childbearing potential and healthy males aged ≥18 and ≤60 years at the time of the screening visit.
* BMI ≥ 18.5 and ≤ 30.0 at the time of the screening visit, and body weight of ≥50 and ≤100 kg.
* Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, ECG and laboratory values at the time of the screening visit, as judged by the Investigator.
* Male participants must be willing to use condom or be vasectomised or practice sexual abstinence from heterosexual intercourse and refrain from donating sperm from the administration of investigational medicinal product (IMP) until 3 months after the administration of IMP. Any female partner of a non-vasectomised male participant who is of child-bearing potential must use a highly effective method of contraception with a failure rate of <1 % to prevent pregnancy from at least 2 weeks prior to the administration of IMP to 3 months after the administration of IMP.
* Women of non-childbearing potential.
* Adequate renal function at the screening visit: Creatinine estimated glomerular filtration rate (eGFR) ≥80 mL/min/1.73 m2 for participants aged 18-50 years and eGFR ≥60 mL/min/1.73 m2 for participants ≥51 years and S-creatinine ≤ upper limit of normal.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial.
* History of kidney disease or renal stone.
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the administration of IMP.
* Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
* Any planned major surgery within the duration of the trial.
* After 10 minutes supine rest at the screening visit, any vital signs values outside the following ranges:

  * Systolic blood pressure: <90 or ≥140 mmHg, or
  * Diastolic blood pressure <50 or ≥90 mmHg, or
  * Pulse <40 or >90 bpm
* A mean QTcF (QT corrected for heart rate by Fredericia's formula) interval of >450 ms after triplicate measurements. The average of the 3 QTc(F) values will be used to determine the participant's eligibility.
* 12-lead ECG:

  * with PR interval shortening < 120 ms.
  * PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre- excitation OR
  * PR interval prolongation > 220 ms OR
  * Intermittent second or third degree atrioventricular (AV) block, or AV dissociation
* History of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome.
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to APC148.
* Regular use of any prescribed or non-prescribed medications, including antacids, analgesics, herbal remedies, vitamins and minerals, within 2 weeks prior to the administration of IMP, except occasional intake of paracetamol (maximum 2000 mg/day and not exceeding 3000 mg/week), as well as nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
* Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis B/C antibodies and/or HIV.
* Positive result for drugs of abuse or alcohol at the screening visit or on admission to the trial site prior to the administration of the IMP.
* Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Participants consented and screened but not dosed in previous Phase I trials are not to be excluded.
* Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times/week is allowed before the screening visit.
* History of, or current, drug abuse, use of anabolic steroids, alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
* Excessive caffeine consumption defined by a daily intake of > 5 cups (1 cup = approximately 240 mL) of caffeine containing beverages, as judged by the Investigator.
* Plasma donation within 1 month of the IMP infusion or blood donation (or corresponding blood loss) during the last 3 months prior to the IMP infusion.
* Participated in a previous cohort in the trial.
* The Investigator considers the participant unlikely to comply with trial procedures, restrictions, and requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Incidence and intensity of adverse events (AEs) | From start of infusion until end of trial visit Day 8
  Frequency, intensity and seriousness of adverse events (AEs) will be assessed. The intensity grades is defined as mild, moderate or severe. AEs will be assessed as not related, possibly or probably related to the investigational medicinal product (IMP)
Incidence and intensity of serious adverse events (SAEs) | From start of infusion until end of trial visit Day 8
  Frequency, intensity and seriousness of Serious adverse events (SAEs) will be assessed. Assessment of causal relationship to IMP will be assessed.
Incidence and intensity of infusion-related AEs | From start of infusion until end of trial visit Day 8
  Frequency, intensity and seriousness of infusion-related adverse events (AEs) will be assessed. The intensity grades is defined as mild, moderate or severe. AEs will be assessed as not related, possibly or probably related to the investigational medicinal product (IMP)
Time course of local tolerability reactions | Pre-dose, Day 1, Day 2 and Day 8
  The infusion site area will be visually inspected before, during and after the IMP infusion. The assessment will include the Investigator's evaluation of swelling, haematoma, and erythema. In addition, each participant will assess their subjective experience of pain and pruritus. Local tolerability reactions will be recorded as infusion-related Adverse events (AEs)
Changes from baseline in blood pressure | Day -1, Day 1, Day 2, Day 3 and Day 8
  Systolic and diastolic blood pressure and pulse will be measured in supine position after 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in respiratory rate | Day -1, Day 1, Day 2, Day 3 and Day 8
  Respiratory rate will be measured in supine position after 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in body temperature | Day1, Day 2, Day 3 and Day 8
  Body temperature will be measured in supine position after 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in heart rate | Day -1, Day 1, Day 2, Day 3 and Day 8
  Heart rate will be measured in supine position after 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in PQ/PR interval | Day -1, Day 1, Day 2, Day 3 and Day 8
  Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. PQ/PR intervals will be recorded. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in QRS interval | Day -1, Day 1, Day 2, Day 3 and Day 8
  Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. QRS intervals will be recorded. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in QT interval | Day -1, Day 1, Day 2, Day 3 and Day 8
  Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. QT intervals will be recorded. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in QTcF interval | Day -1, Day 1, Day 2, Day 3 and Day 8
  Single 12-lead ECG will be recorded in supine position after 10 minutes of rest using an ECG machine. QTcF intervals will be recorded. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in Clinical Laboratory Profile | Day -1, Day 1, Day 2, Day 3 and Day 8
  Safety laboratory data, Clinical chemistry, haematology, and coagulation, will be measured. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator.
Changes from baseline in physical examination | Day -1, Day 1, Day 3 and Day 8
  Assessment of different organ systems. Clinically significant and non-clinically significant abnormal findings will be summarised by treatment and dose.

SECONDARY OUTCOMES:
APC148 plasma concentrations | Day 1, Day 2 and Day 3
  Concentration of APC148 in plasma. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
APC148 urine concentrations | Day 1 and Day 2
  Concentration of APC148 in urine. Urine samples for the determination of plasma concentrations will be collected.
Pharmacokinetic (PK) parameter in plasma - Area under curve (AUC) 0-24 | Day 1, Day 2, Day 3
  Area under the plasma concentration vs. time curve from time 0 to 24 hours. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - AUC0-inf | Day 1, Day 2, Day 3
  AUC from time 0 to infinity. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - AUC0-last | Day 1, Day 2, Day 3
  AUC from time 0 to the last measurable concentration. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - Cmax | Day 1, Day 2, Day 3
  Maximum observed plasma concentration. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - Tmax | Day 1, Day 2, Day 3
  Time to Cmax. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - T1/2 | Day 1, Day 2, Day 3
  Terminal elimination half-life. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - Clearance (CL) | Day 1, Day 2, Day 3
  Total clearance. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - Vz | Day 1, Day 2, Day 3
  Volume of distribution. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameter in plasma - Vss determination of plasma concentrations will be collected. | Day 1, Day 2, Day 3
  Apparent volume of distribution at equilibrium. Venous blood samples (approximately 4 mL) for the determination of plasma concentrations will be collected.
PK parameters in urine - A(e) | Day 1 and Day 2
  Urine samples for the amount of unchanged drug excreted into urine (Ae) will be collected.
PK parameters in urine - fe | Day 1 and Day 2
  Urine samples for the Fraction of IV administered drug that is excreted into urine will be collected.
PK parameter in urine - renal clearance (CLr) | Day 1 and Day 2
  Urine samples for Renal clearance will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Rein-Hedin, MD, Principal Investigator — Clinical Trial Consultants AB (CTC)
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No